CLINICAL TRIAL: NCT02302703
Title: Low FODMAP (Fermentable Oligo-,di-,Mono-saccharides and Polyols) Versus Gluten-free Diet in Pediatric IBS Patients; a Cross-over Randomized Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: fodmap1-HMO-CTIL
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2014-11

CONDITIONS: Effects of Low FODMAP Diet Versus Gluten-free Diet on IBS Symptoms in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the low FODMAP diet (Active Comparator)
  Interventions: Other: low FODMAP diet vs Gluten free diet
- Gluten free diet (Active Comparator)
  Interventions: Other: low FODMAP diet vs Gluten free diet

INTERVENTIONS:
Other: low FODMAP diet vs Gluten free diet

SUMMARY:
Background: IBS (irritable bowel syndrome) describes chronic abdominal pain, which may be relieved with defecation and a change in stool frequency and consistency. Its prevalence among children and adolescents is estimated to be 10-15%. Non-Celiac Gluten Sensitivity is defined as gastrointestinal symptoms which increase with eating gluten-containing foods and improve with a gluten-free diet. FODMAP (fermentable oligo-,di-,mono-saccharides and polyols) are carbohydrates that are not absorbed well in the small intestines, therefore fermented by gut microbiota, increasing osmotic load at the intestine causing fluid shift and gas production. The patient suffers bloating, abdominal pain, flatulence and change of stool consistency. Many foods are FODMAP-rich, including fruit and vegetables, legumes, artificial sweeteners and soft drinks.

Working hypothesis and aims: To study the effect of Low FODMAP diet vs. Gluten free on gastrointestinal symptoms in children with IBS, assuming a beneficial effect based on research in adults.

Methods: 40 children with IBS, aged 6-18 years, will be examined by the pediatric gastroenterology team at Hadassah. All children will record one week of baseline diet and symptoms, then will be randomly selected into a low-FODMAP or Gluten-free diet for one week, together with a washout period of one week between the diets. During the two weeks of intervention diets, the children aided by their parents will document and score symptoms (bowel movements, abdominal pain, flatulence). An analysis of the symptom score will measure the anticipated influence of each diet against baseline diet and symptoms.

Expected results: In previous studies, a change in symptoms was viewed within a few days. We expect to see a reduction of symptoms in one or other of the diets, to prove our hypothesis.

DETAILED DESCRIPTION:
Outline of Study Design, including Plan of the Study and Methods:

Aims: comparing the effects of low FODMAP diet versus gluten-free diet on IBS symptoms in children.

Study design: prospective randomized, crossover trial. Study Population: we are aiming to recruit 40 children aged 6-18 years who answer the pediatric ROME III criteria for IBS. Children will be recruited to the study by physicians at pediatric gastroenterology clinics.

Exclusion criteria:

1. Other diagnosis (e.g. inflammatory bowel disease, celiac disease).
2. Patient receiving chronic medical therapy.
3. Patient already on a restrictive diet (e.g. gluten-free, lactose-free) All patients will document baseline diet - a diary of 7 days by parents/patient specifying exact contents of meals. They will document and score baseline symptoms including stool consistency and frequency, abdominal pain, bloating and flatulence. The baseline documentation will be performed by the child, or by his parents, according to the patient's age and ability.

The patients will be randomly selected to one of the intervention groups. A clinical dietitian has created interventional diets. Half of the patients will start with the low FODMAP diet and half will start with Gluten free. After 7 days, the participants will return to a 7 days washout period of their regular diet. After this period, the groups will switch between the intervention diets, for additional 7 days. During the two weeks of intervention diets, the patients will document and score symptoms as described for the baseline documentation.

-There will be special consideration to several dietary elements in the baseline diet, e.g. patients who may regularly consume high lactose, gluten or FODMAP in their daily diet.

ELIGIBILITY:
Inclusion Criteria:

* children who answer the pediatric ROME III criteria for IBS

Exclusion Criteria:

* Other diagnosis (e.g. inflammatory bowel disease, celiac disease).
* Patient receiving chronic medical therapy.
* Patient already on a restrictive diet (e.g. gluten-free, lactose-free)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-01

PRIMARY OUTCOMES:
abdominal pain score | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel